CLINICAL TRIAL: NCT05635409
Title: STEM-PD Trial: A Multicentre, Single Arm, First in Human, Dose-escalation Trial, Investigating the Safety and Tolerability of Intraputamenal Transplantation of Human Embryonic Stem Cell Derived Dopaminergic Cells for Parkinson's Disease (STEM-PD Product)
Brief Title: A Trial to Determine the Safety and Tolerability of Transplanted Stem Cell Derived Dopamine Neurons to the Brains of Individuals With Parkinson's Disease
Acronym: STEM-PD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCTU0263; 2021-001366-38 (EudraCT Number)
Record Dates: First submitted 2021-11-15; First posted 2022-12-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a multicentre, single arm, dose escalation, first in human advanced therapy investigational medicinal product (ATIMP) trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): The starting dose of this trial is selected as a dose of cells that is likely to be the minimal therapeutic dose, i.e. 100,000 surviving DA neurons per putamen, obtained by transplanting 3.54 million STEM-PD cells per putamen.
  Interventions: Biological: STEM-PD
- Dose 2 (Experimental): To ensure that the investigators are not using a potentially suboptimal cell dose, the investigators also plan to test a higher dose, which is double the dose of dose 1, i.e., 200,000 surviving DA neurons (= 7.08 million transplanted STEM-PD cells) per putamen.
  The Data and Safety Monitoring Board (DSMB) for the trial will make a recommendation for the dosing once participants 1-4 have been dosed and data is available for imaging and clinical measurements, as well as safety reports, 6 months after the last patient has been grafted. The DSMB can recommend either to: i) remain at dose 1; ii) proceed to dose 2; or, iii) wait longer to collect more data. The final decision will be made by the clinical sub-group of the Trial Management Group, after receiving confirmation of the DSMB's recommendation.
  Interventions: Biological: STEM-PD

INTERVENTIONS:
Biological: STEM-PD — STEM-PD is a cryopreserved cell product, consisting of ventral midbrain dopaminergic progenitor cells derived from the clinical-grade hESC line RC17. STEM-PD will be administered using a non-CE marked class III neurosurgical medical device, the Rehncrona-Legradi device, bilaterally in one surgical session to the putamen.

SUMMARY:
Parkinson's disease (PD) occurs when an area of the brain begins to lose nerve cells that produce a chemical called dopamine. Dopamine is an important chemical, and one of its functions is that it helps to regulate body movement. The loss of these nerve cells leads to a reduction of dopamine in the brain. Medications used to treat PD temporarily replace this lost dopamine, but they do not repair the underlying disease. One of the most promising PD therapies to date has been the transplantation of dopamine producing cells into the brain. Unlike current treatments, these therapies may be able to repair the damage caused in PD.

In this trial, the investigators will transplant a new stem cell therapy, called the STEM-PD product, into the area of the brain affected in people with PD. These stem cells can develop into many different cell types, including dopamine-producing nerve cells. The investigators will transplant the stem cells using a device that has been previously used for similar transplants in Lund. This is the first time that the STEM-PD product will be given to humans.

The trial aims to assess whether the STEM-PD product is safe to use in people with PD. The investigators will also be looking for preliminary signs of efficacy.

The trial will recruit participants with PD from the UK and Sweden. Eight participants will undergo the STEM-PD product transplant. Participants will receive a single dose of the STEM-PD product. Participants will attend for 25 visits primarily at their local recruiting hospital. For participants from the UK, some of the imaging will be performed at Invicro (London), and the surgery (including some visits before and after) and some imaging will be performed in Lund. All participants will be followed up for 36 months following surgery

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate in the trial
* Diagnosed with PD as defined using Queens Square Brain Bank criteria
* Moderate disease as defined by having Hoehn and Yahr stage 2-3 in OFF state
* Disease duration > 10 years
* Male or female, aged between 50 and 75 years (inclusive)
* Have a significant response to dopamine therapies as judged by the PI or other delegated clinician
* Have symptoms that are not appropriately controlled by existing oral anti-PD medications, as judged by the PI or other delegated clinician
* Ability to travel to Lund for surgery
* Followed up for at least 12 months prior to inclusion in this trial in the TransEUro observational study
* Be fluent in English/Swedish to enable completion of questionnaires as assessed by the PI or other delegated clinician at Cambridge/Lund, respectively
* Be approved by the TMG clinical sub-group for trial participation

Exclusion Criteria:

* Tremor dominant disease, as assessed by the PI or other delegated clinician
* Significant drug induced dyskinesias as defined by a score of > 2 in the Abnormal Involuntary Movement Scale (AIMS) dyskinesias rating scale, in any body part in the ON state
* Ongoing major medical or psychiatric disorders, including depression (MADRS > 20) and psychosis, that make participation unsuitable, as judged by the PI or other delegated clinician
* Any contraindication to neurosurgery
* Unable to be imaged using MRI
* Extensive ventral striatal loss or normal findings on F-DOPA PET at screening
* Significant cognitive impairment indicative of an incipient dementia/established dementia or values consistent with MoCA score of ≤ 24
* Unable to perform normal copying of interlocking pentagons and/or a semantic fluency score for naming animals of less than 20 over 90 seconds
* Other concomitant treatment with neuroleptics (including atypical neuroleptics) and/or cholinesterase inhibitors
* Previous neurosurgery to the brain, or cell or organ transplantation, or recipient of repeated blood transfusions
* Any contraindication to immunosuppressive therapy, prophylactic antibiotics, and/or osteoporosis prophylaxis (refer to STEM-PD Trial Immunosuppressant Manual)
* High levels of pre-formed specific anti-HLA antibodies to the cell product
* Severely reduced TPMT activity (less than half of the lower normal TPMT activity level)
* History of documented severe/significant allergy requiring treatment
* Female who is pregnant or breastfeeding
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks of the screening visit, or is currently enrolled in an interventional investigational trial
* Female of childbearing potential or male unwilling to follow contraception requirements (see protocol section 12.15)
* Any other condition which, in the opinion of the investigator, makes the patient inappropriate for entry into the trial

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The number and nature of adverse events and serious adverse events in the first 12 months following transplantation | 12 months following transplantation
  Adverse events are recorded from the point of participant informed consent and at every trial visit
Absence of space occupying masses on cranial MRI in the first 12 months following transplantation | 12 months following transplantation
  Magnetic resonance imaging (MRI) scans

SECONDARY OUTCOMES:
Changes in clinical effects at 36 months following transplantation compared to baseline; emergence of new neurological features, | 36 months following transplantation
  A physical examination, to include a review of all body systems as per standard practice will be performed to identify any clinical changes. Specifically, any signs of graft-induced dyskinesias (GIDs) will be looked for.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the Montreal Cognitive Assessment (MoCA) | 36 months following transplantation
  The Montreal Cognitive Assessment (MoCA) is a 30-question test of global cognitive function, which evaluates different types of cognitive abilities, including: orientation, short-term memory, executive function, visuospatial ability, language ability, abstraction, animal naming, and attention. The maximum score is 30 and a score of >26 is considered normal. A higher score is considered a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the Hopkins verbal learning task-revised (HVLT-R) | 36 months following transplantation
  The HVLT-R consists of a 12-item word list, composed of four words each from one of three semantic categories to be learned over the course of three immediate recall learning trials. Participants are also required to undergo a delayed recall trial (requiring free recall of any of the words remembered) and a recognition trial (composed of 24 words, including the 12 target words plus 12 false-positives. A point is given for each correct word and a higher score is considered a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using semantic (animal naming) fluency | 36 months following transplantation
  Participants are asked to name as many animals as possible in 90 seconds. One point is scored for admissible response. A higher score considered a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the stroop test | 36 months following transplantation
  The Stroop test is a measure of verbal processing speed and response inhibition, consisting of three timed trials.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the Digit Span test. | 36 months following transplantation
  Participant is read a list of numbers and asked to repeat the numbers back to the assessor. The lists of numbers gradually gets longer until the participant is unable to remember all of the digits. A backwards span assessment is also completed where the participant is asked to repeat the numbers back in a reverse order.
  One point is scores for each verbatim correct repetition. The total Digit Span total score is a sum of all the forwards and backward scores. A higher score is a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the Boston naming task. | 36 months following transplantation
  In the Boston naming task participants are shown a number of images and are asked to say what the image is. This protocol uses a shortened 15-item version (Lansing et al., 1999) designed for use in patients with neurodegenerative disease. One point for every correct response.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the Wechsler Adult Intelligence Scale (WAIS) similarities test | 36 months following transplantation
  The WAIS similarities assessment includes 14 pairs of words, where participants are asked to name how they are alike or similar. Tests are scored out of 28 and a higher score is considered a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; global cognitive changes assessed using the pentagon copying test | 36 months following transplantation
  In the pentagon copying assessment, participants are asked to copy an intersecting double pentagon figure. Attempts are scored out of a maximum of two points and a higher score is considered a better outcome.
Changes in clinical effects at 36 months following transplantation compared to baseline; changes in non-motor and QOL assessments using the Parkinson's Disease Questionnaire 39 (PDQ-39) | 36 months following transplantation
  The PDQ-39 is a self-rated questionnaire designed to measure PD-related quality of life. It contains 39 questions, covering 8 aspects of quality of life: mobility, activities of daily living (ADL), emotions, stigma, social support, cognition, communication and bodily discomfort. It will be completed by the participant. The total score can be summarised as a percentage, with the score ranging between 0 and 100. A lower scores indicate better health related quality of life.
Changes in clinical effects at 36 months following transplantation compared to baseline; changes in non-motor and QOL assessments using the EuroQol five-dimension, 5 level scale (EQ-5D-5L) | 36 months following transplantation
  The EuroQol five-dimension, 5 level scale (EQ-5D-5L) is a standardised instrument for measuring generic health status in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It will be completed by the participant.
  The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status
Changes in clinical effects at 36 months following transplantation compared to baseline; changes in non-motor and QOL assessments using the PD non motor symptom scale (NMSS). | 36 months following transplantation
  The PD NMSS is a 30-point validated scale which is designed to quantify the extent and severity of non-motor symptoms of PD experienced by the patient. It will be completed by the delegated members of the local research team. Higher scores indicate higher severity and frequency of non-motor symptoms.
Changes in motor features in the OFF state using the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  This is a scale which has sections to be completed by the person with PD together with their carers (if appropriate), as well as sections to be completed by the clinician. Part I assesses the non-motor aspects of experiences of daily living in the week prior to the visit. Part II assesses the motor aspects of experiences of daily living in the week prior to the visit. Part III assesses the motor examination of a participant at the time of the visit (including the Hoehn and Yahr stage), and part IV assesses motor complications in the week prior to the visit. Each item will receive a score ranging from 0 to 4, where 0 represents the absence of impairment and 4 represents the highest degree of impairment.
Changes in motor features in the OFF state using the nine-hole peg test | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The nine-hole peg test is used to measure finger dexterity in participants with neurological diagnoses. It is administered by asking the participant to take the pegs from a container, one by one, and placing them into the holes on the board as quickly as possible. Participants must then remove the pegs, one by one, and replace them into the container. Scores are based on the time taken to complete the test activity.
Changes in motor features in the OFF state using the timed sit-stand-walk test | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The timed sit-stand-walk test is used as a measure of lower extremity strength and speed of walking. Participants begin the test sitting in a chair and told to come to a full stand, then walk 6 metres to a defined point, return to the chair and sit down. The time taken to complete this is measured.
Changes in motor features in the OFF state using the Hauser patient diary card | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The Hauser patient diary card is a 24-hour diary, divided into 30-minute sections. This is used to record PD symptoms and how much time is spent in the different motor states (ON without dyskinesia, ON with non-troublesome dyskinesias, ON with troublesome dyskinesias, OFF, or asleep). Participants will be provided with the diary cards prior to attending the visits and asked to complete this for 3 consecutive days. The completed diary cards will then be collected at the relevant visits.
Changes in motor features in the OFF state using Parkinson KinetiGraph® (PKG®) | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The PKG® is a wrist worn accelerometer from Global Kinetics Pty Ltd. The PKG® watch is worn on the most affected side of the body. Registration will be done for 7 consecutive days just before a visit. For the purposes of this trial, the following data will be collected: bradykinesia and dyskinesia index, OFF time (to correlate with the Hauser patient diary card), and registration of intake of anti-PD medications. Participants will be provided with the PKG® prior to attending the visits to complete data collection and will be asked to return the PKG® at the relevant visit.
  Once the electronic data is transferred from the device to a computer platform, it is processed to generate data.
Changes in motor features in the OFF state using the RUSH dyskinesia scale | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The RUSH dyskinesia scale is a scale to assess the severity of overall dyskinesias based on interference in activities in daily living, to distinguish chorea from dystonia (the two major types of dyskinesias in PD), and to identify the single most disabling form of dyskinesia. A higher score is considered a worse outcome.
Changes in motor features in the OFF state using the Abnormal Involuntary Movement Scale (AIMS) | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The AIMS is used to quantify dyskinesias in the arms, legs or head, and trunk, which includes items such as facial behaviours (jaw, facial muscles, tongue and lips), full-body behaviours (upper, lower, and trunk), and incapacitation due to these movements. The items are scored from 0 to 4, where 0 is normal/healthy and 4 is severely affected.
Changes in motor features in the OFF state using the 30 second tap test | 36 months following transplantation
  Specified motor tasks will be performed in both ON and OFF states. For the OFF state, participants will be asked to stop medication at least 12 hours prior to the visit (for L-dopa/COMT inhibitors) or at least 24 hours (for long-acting dopamine agonists/MAO-B inhibitors).
  The 30 second tap test is a dexterity assessment where the participant is asked to finger tap for 30 seconds. It is tested on both sides, as quickly as possible with the fingers fully open. The number of taps over 30 seconds is registered and the test is performed twice on each hand.
Changes in motor features in the OFF state using a challenge test of levodopa | 36 months following transplantation
  A challenge dose of L-dopa is given, calculated as the participant's average dose (total 24 hours LED/number of dosages per 24 hour period - up to a maximum of 250 mg of L-dopa).
  The challenge dose is given after being off standard L-dopa/COMT inhibitors medications for at least 12 hours or at least 24 hours for long-acting dopamine agonists or L-Dopa preparations and for MAO-B inhibitors, i.e. "practically defined OFF phase". Participants are tested after a low protein breakfast, examples of which will be provided to the participants. After taking the challenge dose, participants will wait for 30 minutes and then perform the MDS-UPDRS part III and the AIMS. These two assessments will then be repeated every 30 minutes up to 120 minutes after taking the challenge dose (or longer if needed, until the L-dopa effect has worn off).
Change in anti-Parkinson medication as measured by change L-dopa equivalent dose | 36 months following transplantation
  At every visit during the trial, a review of concomitant medication (including anti-PD medication) will be performed and any changes recorded. Anti-PD medication will be recorded as a LED, and the change in LED will be monitored throughout the trial.
Changes in F-DOPA uptake and dopamine transporter (DAT) binding at 36 months on PET imaging with F-DOPA and PE2i compared to PET imaging performed pre-transplant | 36 months following transplantation
  The screening F-DOPA PET scans will act as the 'baseline' measurement for changes in F-DOPA uptake. The baseline PE2i will act as the 'baseline' measurement for DAT binding. Changes from this baseline measurement up to and including the 36 months post-transplant time point will be recorded.
The number and nature of SAEs and AEs in the 12 to 36 months period following transplantation | 12 to 36 months period following transplantation
  Adverse events are recorded from the point of participant informed consent and at every trial visit. The difference between this and the primary outcome is that this specifically relates to any safety events reported after the 12 months posttransplant time point.

OTHER OUTCOMES:
Exploratory outcome: changes in F-DOPA uptake and dopamine transporter (DAT) binding at 6 months post transplantation on PET imaging with F-DOPA and PE2i compared to PET imaging performed pre-transplant. | 6 months post transplant
  PET imaging is used within the trial to allow for the assessment of the survival of dopaminergic neurons derived from the transplanted STEM-PD product. The proposed PET ligands to be used within the trial are: F-DOPA, which measures DA synthesis/storage capacity of the transplant, and PE2i, which selectively labels mature DA nerve terminals.
  Positron Emission Tomography (PET) scans are performed with participants in a "practically defined OFF phase".
Exploratory outcome: changes in F-DOPA uptake and dopamine transporter (DAT) binding at 12 months post transplantation on PET imaging with F-DOPA and PE2i compared to PET imaging performed pre-transplant. | 12 months post transplant
  PET imaging is used within the trial to allow for the assessment of the survival of dopaminergic neurons derived from the transplanted STEM-PD product. The proposed PET ligands to be used within the trial are: F-DOPA, which measures DA synthesis/storage capacity of the transplant, and PE2i, which selectively labels mature DA nerve terminals.
  Positron Emission Tomography (PET) scans are performed with participants in a "practically defined OFF phase".
Exploratory outcome: changes in F-DOPA uptake and dopamine transporter (DAT) binding at 24 months post transplantation on PET imaging with F-DOPA and PE2i compared to PET imaging performed pre-transplant. | 24 months post transplant
  PET imaging is used within the trial to allow for the assessment of the survival of dopaminergic neurons derived from the transplanted STEM-PD product. The proposed PET ligands to be used within the trial are: F-DOPA, which measures DA synthesis/storage capacity of the transplant, and PE2i, which selectively labels mature DA nerve terminals.
  Positron Emission Tomography (PET) scans are performed with participants in a "practically defined OFF phase".
Exploratory outcome: change in Fluctuation Dyskinesia Score (FDS) compared to baseline as determined by measurement using wearable movement monitoring devices (Parkinson KinetiGraph™ [PKG]) | 36 months post transplant
  Fluctuation Dyskinesia Score (FDS) is measured using the PKG®, a wrist worn accelerometer from Global Kinetics Pty Ltd. The PKG® watch is worn on the most affected side of the body (same side for all tests). Registration will be done for 7 consecutive days just before a visit. Fluctuation score produced by summing the interquartile range of bradykinesia scores and dyskinesia scores produced very 2 minutes between 09:00-18:00 and expressed as an algorithm. Higher scores are associated with increasing duration of disease, higher levels of medication induced dyskinesia and overall greater degree of symptom variability from dose-to-dose and day-to-day.
Exploratory outcome: change in Dyskinesia score (DKS) compared to baseline as determined by measurement using wearable movement monitoring devices | 36 months post transplant
  Dyskinesia score (DKS) is measured using the PKG®, a wrist worn accelerometer from Global Kinetics Pty Ltd. The PKG® watch is worn on the most affected side of the body (same side for all tests). Registration will be done for 7 consecutive days just before a visit. A higher score is considered a worse outcome.
Exploratory outcome: change in Bradykinesia score (BKS) features compared to baseline as determined by measurement using wearable movement monitoring devices | 36 months post transplant
  Bradykinesia score (BKS) are measured using the PKG®, a wrist worn accelerometer from Global Kinetics Pty Ltd. The PKG® watch is worn on the most affected side of the body (same side for all tests). Registration will be done for 7 consecutive days just before a visit. A higher score is considered a worse outcome.
Levels of donor cell specific anti-human leukocyte antigen (HLA) class I antibodies post-transplant | 36 months post transplant
  HLA antibodies will be monitored throughout the course of the trial via blood tests
Exploratory outcome: changes in markers of inflammation in the cerebrospinal fluid (CSF) | 18 months post transplant
  Optional lumbar punctures will be performed for participants who consented to these. Parameters measured will be decided by the research site and may include routine parameters such as cell count, protein and glucose levels, and presence of oligoclonal bands of immunoglobulins.
Exploratory outcome: change in response to a L-dopa challenge test including measuring the duration and profile of the L-dopa effects between baseline and 36 months: change in MDS-UPDRS Part III score | 36 months post transplant
  For the L-dopa challenge test, participants are given a challenge dose of L-dopa when they are in a practically defined OFF phase. Participants will then perform the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III every 30 minutes for up to 120 minutes. A higher score is considered a worse outcome.
Exploratory outcome: change in response to a L-dopa challenge test including measuring the duration and profile of the L-dopa effects between baseline and 36 months; change in AIMS score | 36 months post transplant
  For the L-dopa challenge test, participants are given a challenge dose of L-dopa when they are in a practically defined OFF phase. Participants will then perform the Abnormal Involuntary Movement Scale (AIMS) every 30 minutes for up to 120 minutes. A higher score is considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Barker, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust & University of Cambridge
Locations (2):
- Region Skåne - Skåne University Hospital, Lund, Sweden
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Summary data will be made available via ClinicalTrials.gov within 1 year of the study's conclusion.
  Individual participant data that underlie results in a publication will be made available with a publication to the extent that it is not expected to lead to identification of individual participants. The nature of the study (a first in human trial with a small number of participants and attention given to the study in the media) means that only limited individual data can be shared without identifying participants.
  Requests for individual data other than those that underlie results in a publication can be sent to the registered trial contact together with a motivation and plan for use of the data. The request will be evaluated by the team.

REFERENCES:
- [Background] Adler AF, Cardoso T, Nolbrant S, Mattsson B, Hoban DB, Jarl U, Wahlestedt JN, Grealish S, Bjorklund A, Parmar M. hESC-Derived Dopaminergic Transplants Integrate into Basal Ganglia Circuitry in a Preclinical Model of Parkinson's Disease. Cell Rep. 2019 Sep 24;28(13):3462-3473.e5. doi: 10.1016/j.celrep.2019.08.058. PMID 31553914
- [Background] Aldrin-Kirk P, Heuer A, Wang G, Mattsson B, Lundblad M, Parmar M, Bjorklund T. DREADD Modulation of Transplanted DA Neurons Reveals a Novel Parkinsonian Dyskinesia Mechanism Mediated by the Serotonin 5-HT6 Receptor. Neuron. 2016 Jun 1;90(5):955-68. doi: 10.1016/j.neuron.2016.04.017. Epub 2016 May 5. PMID 27161524
- [Background] Barker RA, Barrett J, Mason SL, Bjorklund A. Fetal dopaminergic transplantation trials and the future of neural grafting in Parkinson's disease. Lancet Neurol. 2013 Jan;12(1):84-91. doi: 10.1016/S1474-4422(12)70295-8. PMID 23237903
- [Background] Barker RA; TRANSEURO consortium. Designing stem-cell-based dopamine cell replacement trials for Parkinson's disease. Nat Med. 2019 Jul;25(7):1045-1053. doi: 10.1038/s41591-019-0507-2. Epub 2019 Jul 1. PMID 31263283
- [Background] Barker RA, Foltynie T. The future challenges in Parkinson's disease. J Neurol. 2004 Mar;251(3):361-5. doi: 10.1007/s00415-004-0320-8. No abstract available. PMID 15015024
- [Background] Barker RA, Parmar M, Studer L, Takahashi J. Human Trials of Stem Cell-Derived Dopamine Neurons for Parkinson's Disease: Dawn of a New Era. Cell Stem Cell. 2017 Nov 2;21(5):569-573. doi: 10.1016/j.stem.2017.09.014. PMID 29100010
- [Background] Braak H, Bohl JR, Muller CM, Rub U, de Vos RA, Del Tredici K. Stanley Fahn Lecture 2005: The staging procedure for the inclusion body pathology associated with sporadic Parkinson's disease reconsidered. Mov Disord. 2006 Dec;21(12):2042-51. doi: 10.1002/mds.21065. PMID 17078043
- [Background] Braak H, Ghebremedhin E, Rub U, Bratzke H, Del Tredici K. Stages in the development of Parkinson's disease-related pathology. Cell Tissue Res. 2004 Oct;318(1):121-34. doi: 10.1007/s00441-004-0956-9. Epub 2004 Aug 24. PMID 15338272
- [Background] Brundin P, Pogarell O, Hagell P, Piccini P, Widner H, Schrag A, Kupsch A, Crabb L, Odin P, Gustavii B, Bjorklund A, Brooks DJ, Marsden CD, Oertel WH, Quinn NP, Rehncrona S, Lindvall O. Bilateral caudate and putamen grafts of embryonic mesencephalic tissue treated with lazaroids in Parkinson's disease. Brain. 2000 Jul;123 ( Pt 7):1380-90. doi: 10.1093/brain/123.7.1380. PMID 10869050
- [Background] Cardoso T, Adler AF, Mattsson B, Hoban DB, Nolbrant S, Wahlestedt JN, Kirkeby A, Grealish S, Bjorklund A, Parmar M. Target-specific forebrain projections and appropriate synaptic inputs of hESC-derived dopamine neurons grafted to the midbrain of parkinsonian rats. J Comp Neurol. 2018 Sep 1;526(13):2133-2146. doi: 10.1002/cne.24500. Epub 2018 Jul 31. PMID 30007046
- [Background] Defer GL, Geny C, Ricolfi F, Fenelon G, Monfort JC, Remy P, Villafane G, Jeny R, Samson Y, Keravel Y, Gaston A, Degos JD, Peschanski M, Cesaro P, Nguyen JP. Long-term outcome of unilaterally transplanted parkinsonian patients. I. Clinical approach. Brain. 1996 Feb;119 ( Pt 1):41-50. doi: 10.1093/brain/119.1.41. PMID 8624693
- [Background] Evans JR, Barker RA. Neurotrophic factors as a therapeutic target for Parkinson's disease. Expert Opin Ther Targets. 2008 Apr;12(4):437-47. doi: 10.1517/14728222.12.4.437. PMID 18348680
- [Background] Freed CR, Breeze RE, Rosenberg NL, Schneck SA, Kriek E, Qi JX, Lone T, Zhang YB, Snyder JA, Wells TH, et al. Survival of implanted fetal dopamine cells and neurologic improvement 12 to 46 months after transplantation for Parkinson's disease. N Engl J Med. 1992 Nov 26;327(22):1549-55. doi: 10.1056/NEJM199211263272202. PMID 1435881
- [Background] Freed CR, Greene PE, Breeze RE, Tsai WY, DuMouchel W, Kao R, Dillon S, Winfield H, Culver S, Trojanowski JQ, Eidelberg D, Fahn S. Transplantation of embryonic dopamine neurons for severe Parkinson's disease. N Engl J Med. 2001 Mar 8;344(10):710-9. doi: 10.1056/NEJM200103083441002. PMID 11236774
- [Background] Grealish S, Heuer A, Cardoso T, Kirkeby A, Jonsson M, Johansson J, Bjorklund A, Jakobsson J, Parmar M. Monosynaptic Tracing using Modified Rabies Virus Reveals Early and Extensive Circuit Integration of Human Embryonic Stem Cell-Derived Neurons. Stem Cell Reports. 2015 Jun 9;4(6):975-83. doi: 10.1016/j.stemcr.2015.04.011. Epub 2015 May 21. PMID 26004633
- [Background] Hagell P, Piccini P, Bjorklund A, Brundin P, Rehncrona S, Widner H, Crabb L, Pavese N, Oertel WH, Quinn N, Brooks DJ, Lindvall O. Dyskinesias following neural transplantation in Parkinson's disease. Nat Neurosci. 2002 Jul;5(7):627-8. doi: 10.1038/nn863. PMID 12042822
- [Background] Hagell P, Schrag A, Piccini P, Jahanshahi M, Brown R, Rehncrona S, Widner H, Brundin P, Rothwell JC, Odin P, Wenning GK, Morrish P, Gustavii B, Bjorklund A, Brooks DJ, Marsden CD, Quinn NP, Lindvall O. Sequential bilateral transplantation in Parkinson's disease: effects of the second graft. Brain. 1999 Jun;122 ( Pt 6):1121-32. doi: 10.1093/brain/122.6.1121. PMID 10356064
- [Background] Hauser RA, Freeman TB, Snow BJ, Nauert M, Gauger L, Kordower JH, Olanow CW. Long-term evaluation of bilateral fetal nigral transplantation in Parkinson disease. Arch Neurol. 1999 Feb;56(2):179-87. doi: 10.1001/archneur.56.2.179. PMID 10025423
- [Background] Heuer A, Kirkeby A, Pfisterer U, Jonsson ME, Parmar M. hESC-derived neural progenitors prevent xenograft rejection through neonatal desensitisation. Exp Neurol. 2016 Aug;282:78-85. doi: 10.1016/j.expneurol.2016.05.027. Epub 2016 May 25. PMID 27235932
- [Background] Hoban DB, Shrigley S, Mattsson B, Breger LS, Jarl U, Cardoso T, Nelander Wahlestedt J, Luk KC, Bjorklund A, Parmar M. Impact of alpha-synuclein pathology on transplanted hESC-derived dopaminergic neurons in a humanized alpha-synuclein rat model of PD. Proc Natl Acad Sci U S A. 2020 Jun 30;117(26):15209-15220. doi: 10.1073/pnas.2001305117. Epub 2020 Jun 15. PMID 32541058
- [Background] Kefalopoulou Z, Politis M, Piccini P, Mencacci N, Bhatia K, Jahanshahi M, Widner H, Rehncrona S, Brundin P, Bjorklund A, Lindvall O, Limousin P, Quinn N, Foltynie T. Long-term clinical outcome of fetal cell transplantation for Parkinson disease: two case reports. JAMA Neurol. 2014 Jan;71(1):83-7. doi: 10.1001/jamaneurol.2013.4749. PMID 24217017
- [Background] Kirkeby A, Grealish S, Wolf DA, Nelander J, Wood J, Lundblad M, Lindvall O, Parmar M. Generation of regionally specified neural progenitors and functional neurons from human embryonic stem cells under defined conditions. Cell Rep. 2012 Jun 28;1(6):703-14. doi: 10.1016/j.celrep.2012.04.009. Epub 2012 May 26. PMID 22813745
- [Background] Kirkeby A, Nolbrant S, Tiklova K, Heuer A, Kee N, Cardoso T, Ottosson DR, Lelos MJ, Rifes P, Dunnett SB, Grealish S, Perlmann T, Parmar M. Predictive Markers Guide Differentiation to Improve Graft Outcome in Clinical Translation of hESC-Based Therapy for Parkinson's Disease. Cell Stem Cell. 2017 Jan 5;20(1):135-148. doi: 10.1016/j.stem.2016.09.004. Epub 2016 Oct 27. PMID 28094017
- [Background] Kriks S, Shim JW, Piao J, Ganat YM, Wakeman DR, Xie Z, Carrillo-Reid L, Auyeung G, Antonacci C, Buch A, Yang L, Beal MF, Surmeier DJ, Kordower JH, Tabar V, Studer L. Dopamine neurons derived from human ES cells efficiently engraft in animal models of Parkinson's disease. Nature. 2011 Nov 6;480(7378):547-51. doi: 10.1038/nature10648. PMID 22056989
- [Background] Lang AE, Lozano AM. Parkinson's disease. First of two parts. N Engl J Med. 1998 Oct 8;339(15):1044-53. doi: 10.1056/NEJM199810083391506. No abstract available. PMID 9761807
- [Background] Lang AE, Lozano AM. Parkinson's disease. Second of two parts. N Engl J Med. 1998 Oct 15;339(16):1130-43. doi: 10.1056/NEJM199810153391607. PMID 9770561
- [Background] Lehnen D, Barral S, Cardoso T, Grealish S, Heuer A, Smiyakin A, Kirkeby A, Kollet J, Cremer H, Parmar M, Bosio A, Knobel S. IAP-Based Cell Sorting Results in Homogeneous Transplantable Dopaminergic Precursor Cells Derived from Human Pluripotent Stem Cells. Stem Cell Reports. 2017 Oct 10;9(4):1207-1220. doi: 10.1016/j.stemcr.2017.08.016. Epub 2017 Sep 21. PMID 28943253
- [Background] Lewis SJ, Caldwell MA, Barker RA. Modern therapeutic approaches in Parkinson's disease. Expert Rev Mol Med. 2003 Mar 28;5(10):1-20. doi: 10.1017/S1462399403006008. PMID 14987395
- [Background] Li JY, Englund E, Holton JL, Soulet D, Hagell P, Lees AJ, Lashley T, Quinn NP, Rehncrona S, Bjorklund A, Widner H, Revesz T, Lindvall O, Brundin P. Lewy bodies in grafted neurons in subjects with Parkinson's disease suggest host-to-graft disease propagation. Nat Med. 2008 May;14(5):501-3. doi: 10.1038/nm1746. Epub 2008 Apr 6. PMID 18391963
- [Background] Li JY, Englund E, Widner H, Rehncrona S, Bjorklund A, Lindvall O, Brundin P. Characterization of Lewy body pathology in 12- and 16-year-old intrastriatal mesencephalic grafts surviving in a patient with Parkinson's disease. Mov Disord. 2010 Jun 15;25(8):1091-6. doi: 10.1002/mds.23012. PMID 20198645
- [Background] Li W, Englund E, Widner H, Mattsson B, van Westen D, Latt J, Rehncrona S, Brundin P, Bjorklund A, Lindvall O, Li JY. Extensive graft-derived dopaminergic innervation is maintained 24 years after transplantation in the degenerating parkinsonian brain. Proc Natl Acad Sci U S A. 2016 Jun 7;113(23):6544-9. doi: 10.1073/pnas.1605245113. Epub 2016 May 2. PMID 27140603
- [Background] Lindvall O, Rehncrona S, Brundin P, Gustavii B, Astedt B, Widner H, Lindholm T, Bjorklund A, Leenders KL, Rothwell JC, Frackowiak R, Marsden D, Johnels B, Steg G, Freedman R, Hoffer BJ, Seiger A, Bygdeman M, Stromberg I, Olson L. Human fetal dopamine neurons grafted into the striatum in two patients with severe Parkinson's disease. A detailed account of methodology and a 6-month follow-up. Arch Neurol. 1989 Jun;46(6):615-31. doi: 10.1001/archneur.1989.00520420033021. PMID 2786405
- [Background] Mendez I, Dagher A, Hong M, Gaudet P, Weerasinghe S, McAlister V, King D, Desrosiers J, Darvesh S, Acorn T, Robertson H. Simultaneous intrastriatal and intranigral fetal dopaminergic grafts in patients with Parkinson disease: a pilot study. Report of three cases. J Neurosurg. 2002 Mar;96(3):589-96. doi: 10.3171/jns.2002.96.3.0589. PMID 11883846
- [Background] Nolbrant S, Heuer A, Parmar M, Kirkeby A. Generation of high-purity human ventral midbrain dopaminergic progenitors for in vitro maturation and intracerebral transplantation. Nat Protoc. 2017 Sep;12(9):1962-1979. doi: 10.1038/nprot.2017.078. Epub 2017 Aug 31. PMID 28858290
- [Background] Olanow CW, Goetz CG, Kordower JH, Stoessl AJ, Sossi V, Brin MF, Shannon KM, Nauert GM, Perl DP, Godbold J, Freeman TB. A double-blind controlled trial of bilateral fetal nigral transplantation in Parkinson's disease. Ann Neurol. 2003 Sep;54(3):403-14. doi: 10.1002/ana.10720. PMID 12953276
- [Background] Palfi S, Gurruchaga JM, Ralph GS, Lepetit H, Lavisse S, Buttery PC, Watts C, Miskin J, Kelleher M, Deeley S, Iwamuro H, Lefaucheur JP, Thiriez C, Fenelon G, Lucas C, Brugieres P, Gabriel I, Abhay K, Drouot X, Tani N, Kas A, Ghaleh B, Le Corvoisier P, Dolphin P, Breen DP, Mason S, Guzman NV, Mazarakis ND, Radcliffe PA, Harrop R, Kingsman SM, Rascol O, Naylor S, Barker RA, Hantraye P, Remy P, Cesaro P, Mitrophanous KA. Long-term safety and tolerability of ProSavin, a lentiviral vector-based gene therapy for Parkinson's disease: a dose escalation, open-label, phase 1/2 trial. Lancet. 2014 Mar 29;383(9923):1138-46. doi: 10.1016/S0140-6736(13)61939-X. Epub 2014 Jan 10. PMID 24412048
- [Background] Schade S, Mollenhauer B, Trenkwalder C. Levodopa Equivalent Dose Conversion Factors: An Updated Proposal Including Opicapone and Safinamide. Mov Disord Clin Pract. 2020 Mar 16;7(3):343-345. doi: 10.1002/mdc3.12921. eCollection 2020 Apr. No abstract available. PMID 32258239
- [Background] Schuepbach WM, Rau J, Knudsen K, Volkmann J, Krack P, Timmermann L, Halbig TD, Hesekamp H, Navarro SM, Meier N, Falk D, Mehdorn M, Paschen S, Maarouf M, Barbe MT, Fink GR, Kupsch A, Gruber D, Schneider GH, Seigneuret E, Kistner A, Chaynes P, Ory-Magne F, Brefel Courbon C, Vesper J, Schnitzler A, Wojtecki L, Houeto JL, Bataille B, Maltete D, Damier P, Raoul S, Sixel-Doering F, Hellwig D, Gharabaghi A, Kruger R, Pinsker MO, Amtage F, Regis JM, Witjas T, Thobois S, Mertens P, Kloss M, Hartmann A, Oertel WH, Post B, Speelman H, Agid Y, Schade-Brittinger C, Deuschl G; EARLYSTIM Study Group. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. 2013 Feb 14;368(7):610-22. doi: 10.1056/NEJMoa1205158. PMID 23406026
- [Background] Schupbach WM, Maltete D, Houeto JL, du Montcel ST, Mallet L, Welter ML, Gargiulo M, Behar C, Bonnet AM, Czernecki V, Pidoux B, Navarro S, Dormont D, Cornu P, Agid Y. Neurosurgery at an earlier stage of Parkinson disease: a randomized, controlled trial. Neurology. 2007 Jan 23;68(4):267-71. doi: 10.1212/01.wnl.0000250253.03919.fb. Epub 2006 Dec 6. PMID 17151341
- [Background] Tiklova K, Nolbrant S, Fiorenzano A, Bjorklund AK, Sharma Y, Heuer A, Gillberg L, Hoban DB, Cardoso T, Adler AF, Birtele M, Lunden-Miguel H, Volakakis N, Kirkeby A, Perlmann T, Parmar M. Single cell transcriptomics identifies stem cell-derived graft composition in a model of Parkinson's disease. Nat Commun. 2020 May 15;11(1):2434. doi: 10.1038/s41467-020-16225-5. PMID 32415072
- [Background] Voon V, Krack P, Lang AE, Lozano AM, Dujardin K, Schupbach M, D'Ambrosia J, Thobois S, Tamma F, Herzog J, Speelman JD, Samanta J, Kubu C, Rossignol H, Poon YY, Saint-Cyr JA, Ardouin C, Moro E. A multicentre study on suicide outcomes following subthalamic stimulation for Parkinson's disease. Brain. 2008 Oct;131(Pt 10):2720-8. doi: 10.1093/brain/awn214. PMID 18941146
- [Background] Wider C, Pollo C, Bloch J, Burkhard PR, Vingerhoets FJ. Long-term outcome of 50 consecutive Parkinson's disease patients treated with subthalamic deep brain stimulation. Parkinsonism Relat Disord. 2008;14(2):114-9. doi: 10.1016/j.parkreldis.2007.06.012. Epub 2007 Sep 5. PMID 17822940
- [Background] Wijeyekoon R, Barker RA. Cell replacement therapy for Parkinson's disease. Biochim Biophys Acta. 2009 Jul;1792(7):688-702. doi: 10.1016/j.bbadis.2008.10.007. Epub 2008 Oct 25. PMID 19007882
- [Background] Witt K, Daniels C, Reiff J, Krack P, Volkmann J, Pinsker MO, Krause M, Tronnier V, Kloss M, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G. Neuropsychological and psychiatric changes after deep brain stimulation for Parkinson's disease: a randomised, multicentre study. Lancet Neurol. 2008 Jul;7(7):605-14. doi: 10.1016/S1474-4422(08)70114-5. Epub 2008 Jun 4. PMID 18538636
- [Background] Lansing AE, Ivnik RJ, Cullum CM, Randolph C. An empirically derived short form of the Boston naming test. Arch Clin Neuropsychol. 1999 Aug;14(6):481-7. PMID 14590575
- [Derived] Paul G, Bjartmarz H, Bjorklund A, Cutting E, Evans A, Harry B, Hansson O, Kayhanian S, Kirkeby A, Lao-Kim N, Lindvall O, Nelander J, Piccini P, Smith R, Ullen S, Van Vliet T, Widner H, Parmar M, Barker RA. STEM-PD trial protocol: a multi-centre, single-arm, first-in-human, dose-escalation trial, investigating the safety and tolerability of intraputamenal transplantation of human embryonic stem cell-derived dopaminergic cells for Parkinson's disease. BMJ Open. 2025 Dec 30;15(12):e107597. doi: 10.1136/bmjopen-2025-107597. PMID 41469040
- See also: World's first clinical trial to treat Parkinson's disease with stem cells — https://sitn.hms.harvard.edu/flash/2018/worlds-first-clinical-trial-treat-parkinsons-disease-stem-cells/
- See also: Surgical instrument for implantation — https://shorturl.at/qZoLQ